CLINICAL TRIAL: NCT03951766
Title: An Online Pilot Study of Version 2 of the Smoking Cessation Smartphone App "Smiling Instead of Smoking" (SiS)
Brief Title: Version 2 of the Smoking Cessation Smartphone App "Smiling Instead of Smoking" (SiS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Bettina B. Hoeppner, Associate Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P002699
Record Dates: First submitted 2019-05-07; First posted 2019-05-15 (Actual); Results first posted 2021-09-09 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Smoking Cessation; Smoking, Tobacco
Keywords: mHealth; smartphone; smoking cessation; app; happiness; positive psychology; nondaily smoking
MeSH Terms: conditions — Smoking Cessation; Tobacco Smoking; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Pilot study: all participants will use the smartphone app for a total of 7 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smiling Instead of Smoking App (Other): This is a pilot study; all participants will use the app in the same manner/time period.
  Interventions: Behavioral: Smiling Instead of Smoking (SiS) App Version 2

INTERVENTIONS:
Behavioral: Smiling Instead of Smoking (SiS) App Version 2 — The investigators have developed a smartphone app that acts as a behavioral, in-the-pocket coach and uses positive psychology exercises to enhance quitting success. It is anonymous, portable, and provides just-in-time support, an important feature for smokers who smoke under specific conditions and circumstances. To support treatment, investigators use a positive psychology approach. The smartphone app administers positive psychology exercises to enhance and/or maintain positive affect, which is hypothesized to stimulate nondaily smokers to enact healthier alternatives to smoking by broadening their thought-action repertoire, increasing confidence, and decreasing craving and defensiveness about smoking-related health information.

SUMMARY:
The overall goal of this pilot study is to solicit feedback from nondaily smokers looking for smoking cessation support online (n=90) about Version 2 of a smartphone app investigators designed to support smoking cessation, and to test if within-person theorized mechanisms of change are occurring as participants undergo the app-assisted quit attempt. Data sources will be passively collected smartphone app usage data, surveys and, in a sub-sample (n=20), online video-conference user feedback sessions. Results will be used to guide the design of Version 3.0 of the "Smiling Instead of Smoking" (SiS) smartphone app. Specifically, the aims of this study are to:

1. Assess ease-of-use and helpfulness of the app, as rated by app users 6 weeks after their chosen smoking cessation date
2. Test if within-person changes occur in theorized mechanisms of behavior change as nondaily smokers undergo a SiS app assisted quit attempt
3. Identify app features in need of improvement, as identified by passively recorded app usage patterns, REDCap open-ended survey items, and, in a sub-sample, user feedback sessions (n=20)

DETAILED DESCRIPTION:
An estimated 90 participants will participate in this study based on the following eligibility criteria: (a) 18+ years of age, (b) smartphone ownership (c) current nondaily smoker, who smokes at least weekly, and no more than 25 out of the past 30 days (i.e., 71% of nondaily smokers), and (d) has current quit intention (i.e., 65-74% of nondaily smokers). Investigators will stop enrollment when n=90 participants have completed the primary endpoint of the study, which is the 6-week follow-up. This study will be conducted entirely remotely and will require a screening process prior to enrolling participants on the app.

Study participation will last 6 months, where surveys will be administered prior to the quit day (online, as part of a screening test), and at 2-week, 6-week, 3-month, and 6-month follow-ups of the participant's chosen quit day. Participants will use the app for a strongly encouraged period of 7 weeks (1 week before, 6 weeks following the quit attempt), and optional continued use thereafter.

Participants will complete two types of assessment: (1) surveys, and (2) (in a sub-sample) user feedback sessions conducted via phone and/or video-conference call. Potential participants will click-through to the study website. This website will explain that participants must call study staff in order to be phone-screened and to participate in the study. During the phone-screen, participants will be directed to complete an online survey via REDCap. If participants complete the survey and pass the screening test (e.g., correctly responding to reading-check items in the online survey), they choose a smoking cessation quit day, and schedule a phone call with study staff to enroll in the study. This enrollment phone call occurs 1 week prior to the chosen quit day. During this call, study staff will provide the link to download the app, and provide participants with an app-walkthrough. Thereafter, participants will receive survey links for 2-week, 6-week, 3-month and 6-month follow-ups via an emailed link.

Participation in the user feedback session is optional. Within the baseline survey, participants will be asked if they would be willing to participate in an online video-conference user feedback session after they have used the app for seven weeks (1 week pre, 6 weeks post their chosen smoking quit day). If selected for the online user feedback sessions (selected at random from interested participants, with stratification based on gender, age, and race/ethnicity), participants will receive an email and/or phone call upon completing their 6-week survey to set up the user feedback session.

The online user feedback sessions (n=20) will consist of the participants, and 1-2 members of the study staff. Relatively little guidance will be provided in this setting. Instead, 4 open-ended questions will be posed (i.e., did the app help you in your quit attempt? What did you like? What did you dislike? How could the app be improved?). All conference calls will be recorded for later analysis.

Sample size and Power Considerations: The primary goal of this study is to gather qualitative input rather than data to detect a pre-specified effect. The goal of this pilot study is to get input from app users who are interacting with the app and study staff completely remotely, without the benefit of in-person interaction, which is closer to the real-world experience potential users would have than the participants in Study 1.

Planned Analyses:

Aim 1 (Ease-of-use and usefulness). To assess the degree to which SiS Version 2 is easy to use and perceived as useful by nondaily smokers attempting to quit smoking, investigators will use the Week 6 survey data, and will calculate means and standard deviations for the survey items querying ease of use and usefulness for each feature of the app.

Aim 2 (Within-person changes). To test if nondaily smokers utilizing SiS Version 2 experienced changes over time on constructs theorized to underlie smoking cessation, investigators will use the online survey data and fit one repeated measures mixed effects model per construct of interest (i.e., desire to smoke, mood, self-efficacy to quit/stay quit, motivation, outcome expectancies such as pros/cons, stress, coping), where the construct will be the dependent variable, and time (0=baseline, 1=2-week, 2=6-week, 3=3-month, 4=6-month) will be the predictor. Correlations over time will be modeled with an unstructured covariance matrix. The primary endpoint is 6 weeks post quit (i.e., end of treatment). A contrast statement will be used to compare baseline versus 6-week follow-up. Given the explorative nature of this study, investigators will not correct for multiple testing.

Aim 3 (Identify app features in need of improvement). To identify features of the app that are in need of improvement, investigators will examine the passively generated app usage data generated by study participants as they undergo their quit attempts, and will generate descriptive summary statistics on these usage data. To gain deeper insight, investigators will also conduct user feedback sessions with a randomly selected subsample of participants.

ELIGIBILITY:
Inclusion Criteria:

* Owns a smartphone
* Is a nondaily smoker, who smokes at least weekly and no more than 25 out of the past 30 days
* Has a current intention to quit smoking
* Interested in using a smartphone app to quit smoking

Exclusion Criteria:

* Under 18 years of age
* Does not own a smartphone
* Is not a nondaily smoker, who smokes at least weekly and no more than 25 out of the past 30 days
* Does not have a current intention to quit smoking
* Is not interested in using a smartphone app to quit smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bettina B Hoeppner, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Investigators do not plan to share IPD with any other researchers.

REFERENCES:
- [Background] Cox LS, Tiffany ST, Christen AG. Evaluation of the brief questionnaire of smoking urges (QSU-brief) in laboratory and clinical settings. Nicotine Tob Res. 2001 Feb;3(1):7-16. doi: 10.1080/14622200020032051. PMID 11260806
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Etter JF, Bergman MM, Humair JP, Perneger TV. Development and validation of a scale measuring self-efficacy of current and former smokers. Addiction. 2000 Jun;95(6):901-13. doi: 10.1046/j.1360-0443.2000.9569017.x. PMID 10946439
- [Background] Etter JF, Humair JP, Bergman MM, Perneger TV. Development and validation of the Attitudes Towards Smoking Scale (ATS-18). Addiction. 2000 Apr;95(4):613-25. doi: 10.1046/j.1360-0443.2000.95461312.x. PMID 10829336
- [Background] Kahler CW, Lachance HR, Strong DR, Ramsey SE, Monti PM, Brown RA. The commitment to quitting smoking scale: initial validation in a smoking cessation trial for heavy social drinkers. Addict Behav. 2007 Oct;32(10):2420-4. doi: 10.1016/j.addbeh.2007.04.002. Epub 2007 Apr 6. PMID 17478057
- [Background] Asher MK, Martin RA, Rohsenow DJ, MacKinnon SV, Traficante R, Monti PM. Perceived barriers to quitting smoking among alcohol dependent patients in treatment. J Subst Abuse Treat. 2003 Mar;24(2):169-74. doi: 10.1016/s0740-5472(02)00354-9. PMID 12745034
- [Background] Ward RM, Velicer WF, Rossi JS, Fava JL, Prochaska JO. Factorial invariance and internal consistency for the decisional balance inventory--short form. Addict Behav. 2004 Jul;29(5):953-8. doi: 10.1016/j.addbeh.2004.02.042. PMID 15219341
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Lyubomirsky, S., & Lepper, H. (1999). A measure of subjective happiness: Preliminary reliability and construct validation. Social Indicators Research, 46, 137-155.
- [Derived] Hoepper BB, Siegel KR, Carlon HA, Kahler CW, Park ER, Taylor ST, Simpson HV, Hoeppner SS. Feature-Level Analysis of a Smoking Cessation Smartphone App Based on a Positive Psychology Approach: Prospective Observational Study. JMIR Form Res. 2022 Jul 28;6(7):e38234. doi: 10.2196/38234. PMID 35900835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between 06/24/2019 and 11/15/2019. Study recruitment information was displayed on Craigslist, Facebook, Reddit, Smokefree.gov, ClinicalTrials.gov, a study recruitment website at Massachusetts General Hospital, our study website, and websites of local universities. Recruitment was bolstered through word of mouth referrals.
Pre-assignment Details: All participants who were enrolled were assigned to the single treatment arm.
Groups:
- Smiling Instead of Smoking App: This is a pilot study; all participants will use the app in the same manner/time period (i.e., this is a single-arm trial)t.
  Smiling Instead of Smoking (SiS) App Version 2: The investigators have developed a smartphone app that acts as a behavioral, in-the-pocket coach and uses positive psychology exercises to enhance quitting success. It is anonymous, portable, and provides just-in-time support, an important feature for smokers who smoke under specific conditions and circumstances. To support treatment, investigators use a positive psychology approach. The smartphone app administers positive psychology exercises to enhance and/or maintain positive affect, which is hypothesized to stimulate nondaily smokers to enact healthier alternatives to smoking by broadening their thought-action repertoire, increasing confidence, and decreasing craving and defensiveness about smoking-related health information.
Period: Treatment Phase
Arm/Group | Smiling Instead of Smoking App
Started | 100
Completed | 99
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Follow-up Phase
Arm/Group | Smiling Instead of Smoking App
Started | 99
Completed | 89
Not Completed | 10
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Groups:
- Smiling Instead of Smoking (SiS) App Version 2: Behavioral: Smiling Instead of Smoking (SiS) App Version 2 The investigators have developed a smartphone app that acts as a behavioral, in-the-pocket coach and uses positive psychology exercises to enhance quitting success. It is anonymous, portable, and provides just-in-time support, an important feature for smokers who smoke under specific conditions and circumstances. To support treatment, investigators use a positive psychology approach. The smartphone app administers positive psychology exercises to enhance and/or maintain positive affect, which is hypothesized to stimulate nondaily smokers to enact healthier alternatives to smoking by broadening their thought-action repertoire, increasing confidence, and decreasing craving and defensiveness about smoking-related health information.
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (11.4)
Sex/Gender, Customized [Count of Participants; unit: Participants] — self-reported gender ("What is your gender?", answer options: male, female, other)
  Participants
    Self-reported gender identity: Female | 61
    Self-reported gender identity: Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 88
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 75
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 100
Number of days smoked in past 30 days [Mean (Standard Deviation); unit: days] | 14.7 (4.6)
Number of cigarettes smoked per smoking day [Mean (Standard Deviation); unit: number of cigarettes per day] | 4.6 (3.3)
Ever smoked daily [Count of Participants; unit: Participants] | 70
Ever quit before [Count of Participants; unit: Participants] | 77

OUTCOME MEASURES:

1. Primary Outcome: Ease-of-use and Helpfulness of the App
Description: As rated by app users 6 weeks after their chosen smoking cessation date via open-ended REDCap survey. This survey asks questions concerning feasibility, usefulness, and overall opinions of specific app features. Responses were rated on 4-point Likert-scales with ease-of-use rated with the options 0 = Not easy at all | 1 = Somewhat easy to use | 2 = Easy to use | 3 = Very easy to use, and usefulness rated with the options 0 = Not at all useful | 1 = Somewhat useful | 2 = Useful | 3 = Very useful. For both ease-of-use and usefulness items, scores range from 0 to 3 with higher scores indicating a better opinion of the app features.
Time Frame: 6 weeks after chosen smoking cessation date
Population: Of the 99 people still active in the trial at the end-of-treatment visit, 4 had missing data for all ease-of-use and helpfulness ratings, and 1-2 people had missing ratings for some but not all items on this questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
Number analyzed (Participants) | 95
units on a scale
  Ease of use: Completing the positive psychology exercises every day. | 2.39 (0.89)
  Ease of use: Specifically, completing the specific exercise called 3 Good Things. | 2.36 (0.89)
  Ease of use: Specifically, completing the specific exercise called Savoring. | 2.42 (0.79)
  Ease of use: Specifically, completing the specific exercise called Experiencing Kindness.: number analyzed (Participants) | 93
  Ease of use: Specifically, completing the specific exercise called Experiencing Kindness. | 2.39 (0.90)
  Ease of use: Specifically, completing the specific exercise called Reliving Happy Moments. | 2.54 (0.77)
  Ease of use: Specifically, completing the specific exercise called Rose, Thorn and Bud. | 2.40 (0.83)
  Ease of use: Viewing your past happiness exercises in the Happiness Log. | 2.64 (0.67)
  Ease of use: Viewing Owl Wisdoms within the Treasure Chest menu. | 2.57 (0.65)
  Ease of use: Setting and re-setting your quit day. | 2.51 (0.77)
  Ease of use: Completing the behavioral challenges. | 2.52 (0.73)
  Ease of use: Accessing and updating your cigarette log. | 2.61 (0.75)
  Ease of use: Accessing the I have a craving feature (Magma Bear game).: number analyzed (Participants) | 94
  Ease of use: Accessing the I have a craving feature (Magma Bear game). | 2.32 (0.94)
  Ease of use: Adding and being reminded of your smoke alarms within the Action Plan menu. | 2.37 (0.84)
  Ease of use: Adding and viewing your personal reasons for quitting within the Action Plan menu. | 2.47 (0.78)
  Ease of use: Viewing strategies for remaining smoke-free within the Action Plan menu. | 2.55 (0.68)
  Ease of use: Viewing your earned badges within the Treasure Chest menu. | 2.65 (0.56)
  Ease of use: Viewing benefits of quitting within the Treasure Chest menu. | 2.58 (0.61)
  Usefulness: Completing the positive psychology exercises every day.: number analyzed (Participants) | 94
  Usefulness: Completing the positive psychology exercises every day. | 2.19 (0.90)
  Usefulness: Specifically, completing the specific exercise called 3 Good Things. | 2.23 (0.92)
  Usefulness: Specifically, completing the specific exercise called Savoring. | 2.16 (0.95)
  Usefulness: Specifically, completing the specific exercise called Experiencing Kindness. | 2.13 (0.98)
  Usefulness: Specifically, completing the specific exercise called Reliving Happy Moments. | 2.22 (0.92)
  Usefulness: Specifically, completing the specific exercise called Rose, Thorn and Bud. | 2.09 (0.96)
  Usefulness: Viewing your past happiness exercises within the Happiness Log. | 2.16 (0.90)
  Usefulness: . Viewing Owl Wisdoms within the Treasure Chest menu. | 2.19 (0.91)
  Usefulness: Setting and re-setting your quit day. | 2.07 (0.98)
  Usefulness: Completing the behavioral challenges. | 2.21 (0.90)
  Usefulness: Accessing and updating your cigarette log. | 2.39 (0.82)
  Usefulness: Using the I have a craving feature (Magma Bear game). | 1.32 (1.24)
  Usefulness: Adding and being reminded of your smoke alarms within the Action Plan menu. | 2.08 (0.96)
  Usefulness: Adding and viewing your personal reasons for quitting within the Action Plan menu. | 2.34 (0.82)
  Usefulness: Viewing strategies for remaining smoke-free within the Action Plan menu. | 2.29 (0.86)
  Usefulness: Viewing your earned badges within the Treasure Chest menu.: number analyzed (Participants) | 94
  Usefulness: Viewing your earned badges within the Treasure Chest menu. | 2.01 (1.03)
  Usefulness: Viewing benefits of quitting within the Treasure Chest menu.: number analyzed (Participants) | 94
  Usefulness: Viewing benefits of quitting within the Treasure Chest menu. | 2.21 (0.89)

2. Secondary Outcome: Within-person Changes in Theorized Mechanism of Behavior Change - Questionnaire of Smoking Urges (Cox et al., 2001)
Description: This 10-item scale assesses overall nicotine dependence, craving, and smoking withdrawal symptoms. Items were rated on a 7-point Likert-scale ranging from 1=Strongly disagree to 7=Strongly agree. We presented mean instead of total scores for ease in interpretation, so that scale scores can range from 1.0 to 7.0, with higher scores indicating greater smoking urges.
Time Frame: Baseline, 2-weeks, and 6-weeks post-quit
Population: Some participants had missing data for follow-up time-points. In the statistical analysis, we used hierarchical linear mixed models with maximum likelihood estimation to handle missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Smiling Instead of Smoking (SiS) App Version 2: Behavioral: Smiling Instead of Smoking (SiS) Smartphone App Version 2
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
Number analyzed (Participants) | 100
units on a scale
  Baseline | 3.66 (1.36)
  Week 2: number analyzed (Participants) | 96
  Week 2 | 2.50 (1.38)
  Week 6: number analyzed (Participants) | 95
  Week 6 | 2.18 (1.57)
Statistical Analysis 1: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority; p < .0001, t-test, 2 sided — The a priori threshold for statistical significance was alpha=.05. We did not adjust for multiple comparisons, because this was a secondary outcome. The p-value is for a planned specific comparison of week 6 to baseline; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-1.9 to -1.1]

3. Secondary Outcome: Within-person Changes in Theorized Mechanism of Behavior Change - Single-item Urges Measure
Description: Single-item measure: "Right now, how strong is your desire/urge to smoke?". This single-item measure was rated on a scale of "0, not at all strong" to "100, extremely strong", so that higher scores indicate stronger smoking urges.
Time Frame: Baseline, 2-weeks, and 6-weeks post-quit
Population: n=1 participants were missing baseline data for this survey; n=4 and n=6 participants had missing data at weeks 2 and 6, respectively. Data was analyzed in a hierarchical mixed model with maximum likelihood estimation to handle missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
Number analyzed (Participants) | 99
units on a scale
  Baseline | 50.87 (27.03)
  Week 2: number analyzed (Participants) | 96
  Week 2 | 31.27 (29.31)
  Week 6: number analyzed (Participants) | 94
  Week 6 | 26.12 (30.90)
Statistical Analysis 1: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority; p < .0001, t-test, 2 sided — We used hierarchical linear mixed models with maximum likelihood estimation to handle missing data, then used a planned, pairwise comparison to test for within-person changes between baseline and week 6; Median Difference (Final Values) = -24.9, 95% CI 2-sided [-32.7 to -17.1]

4. Secondary Outcome: Within-person Changes in Theorized Mechanism of Behavior Change - Positive and Negative Affect Schedule (Watson et al., 1988)
Description: This 20-item scale measures positive and negative. Participants were asked to indicate how they felt in the past week, using a 5-point Likert scale ranging from 1="very slightly or not at all" to 5="extremely." Scores for 10 positive words and 10 negative words were summed separately and were reported as mean scores (not scale totals) ranging from 1-5, with lower scores indicating low (positive or negative) affect and higher scores indicating high (positive or negative) affect. The 10 items for POSITIVE (PA) affect are attentive, interested, alert, excited, enthusiastic, inspired, proud, determined, strong, and active. The 10 items for NEGATIVE (NA) affect are distressed, upset, hostile, irritable, scared, afraid, ashamed, guilty, nervous, and jittery.
Time Frame: Baseline, 2-weeks, and 6-weeks post-quit
Population: n=1 had incomplete baseline data, n=6 were missing Week 2 data, n=5 were missing Week 6 data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
Number analyzed (Participants) | 100
units on a scale
  PANAS - Positive Affect - Baseline: number analyzed (Participants) | 99
  PANAS - Positive Affect - Baseline | 3.39 (0.82)
  PANAS - Positive Affect - Week 2: number analyzed (Participants) | 94
  PANAS - Positive Affect - Week 2 | 3.47 (0.77)
  PANAS - Positive Affect - Week 6: number analyzed (Participants) | 95
  PANAS - Positive Affect - Week 6 | 3.59 (0.90)
  PANAS - Negative Affect - Baseline: number analyzed (Participants) | 99
  PANAS - Negative Affect - Baseline | 2.32 (1.02)
  PANAS - Negative Affect - Week 2: number analyzed (Participants) | 95
  PANAS - Negative Affect - Week 2 | 2.13 (0.79)
  PANAS - Negative Affect - Week 6: number analyzed (Participants) | 95
  PANAS - Negative Affect - Week 6 | 2.18 (1.10)
Statistical Analysis 1: Comparison: Smiling Instead of Smoking (SiS) App Version 2; PANAS positive affect; Test type: Superiority; p = 0.06, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.0 to 0.4]
Statistical Analysis 2: Comparison: Smiling Instead of Smoking (SiS) App Version 2; PANAS negative affect; Test type: Superiority; p = 0.36, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.1]

5. Secondary Outcome: Within-person Changes in Theorized Mechanism of Behavior Change - Subjective Happiness Scale (Lyubomirsky & Lepper, 1999)
Description: This 4-item scale assesses global subjective happiness. Each question is rated on a Likert-scale of 1-7. Scale scores were reported as mean scores in this study, with higher scores indicating higher subjective happiness.
Time Frame: Baseline, 2-weeks, and 6-weeks post-quit
Population: n=1 had incomplete baseline data, n=6 were missing Week 2 data, n=5 were missing Week 6 data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
Number analyzed (Participants) | 100
units on a scale
  Baseline | 4.77 (1.39)
  Week 2: number analyzed (Participants) | 96
  Week 2 | 4.81 (1.38)
  Week 6: number analyzed (Participants) | 95
  Week 6 | 4.94 (1.42)
Statistical Analysis 1: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority; p = 0.1627, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.1 to 0.4]

6. Secondary Outcome: Within-person Changes in Theorized Mechanism of Behavior Change - Single-item Happiness Measures
Description: Two single-item happiness measures were used: "In the PAST WEEK, how happy have you felt?" and "How happy are you feeling RIGHT NOW?". Both items were rated on slider scales ranging from 0="not at all" to 100="extremely", such that higher scores indicate greater levels of happiness.
Time Frame: Baseline, 2-weeks, and 6-weeks post-quit
Population: n=1 had incomplete baseline data, n=4 were missing Week 2 data, n=7 were missing Week 6 data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
Number analyzed (Participants) | 99
units on a scale
  Happiness Past Week - Baseline | 67.74 (21.50)
  Happiness Past Week - Week 2: number analyzed (Participants) | 96
  Happiness Past Week - Week 2 | 67.75 (21.88)
  Happiness Past Week - Week 6: number analyzed (Participants) | 93
  Happiness Past Week - Week 6 | 69.69 (23.91)
  Happiness Right Now - Baseline | 70.04 (20.38)
  Happiness Right Now - Week 2: number analyzed (Participants) | 96
  Happiness Right Now - Week 2 | 68.55 (25.34)
  Happiness Right Now - Week 6: number analyzed (Participants) | 95
  Happiness Right Now - Week 6 | 70.03 (24.93)
Statistical Analysis 1: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Single-item - past week; Test type: Superiority; p = 0.62, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-3.8 to 6.3]
Statistical Analysis 2: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Single-item - right now; Test type: Superiority; p = 0.83, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-5.4 to 4.4]

7. Secondary Outcome: Within-person Changes in Theorized Mechanism of Behavior Change - Self-Efficacy to Abstain From Smoking Questionnaire (Etter et al., 2000)
Description: The 12-item Smoking Self-Efficacy Questionnaire (SEQ-12) assesses confidence to abstain from smoking when faced with internal stimuli (6 items; e.g., when I feel very anxious) and external stimuli (6 items; e.g., after a meal). Items were assessed on slider scales ranging from 0="not at all confident" to 100="extremely confident" and results are presented as mean scale scores, where higher scores indicate greater self-efficacy to abstain from smoking.
Time Frame: Baseline, 2-weeks, and 6-weeks post-quit
Population: n=1 had incomplete baseline data, n=4 were missing Week 2 data, n=5 were missing Week 6 data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
Number analyzed (Participants) | 100
units on a scale
  SEQ Internal Cues - Baseline | 53.44 (22.04)
  SEQ Internal Cues - Week 2: number analyzed (Participants) | 96
  SEQ Internal Cues - Week 2 | 60.15 (23.33)
  SEQ Internal Cues - Week 6: number analyzed (Participants) | 95
  SEQ Internal Cues - Week 6 | 66.98 (29.09)
  SEQ External Cues - Baseline | 58.89 (21.10)
  SEQ External Cues - Week 2: number analyzed (Participants) | 96
  SEQ External Cues - Week 2 | 64.75 (23.31)
  SEQ External Cues - Week 6: number analyzed (Participants) | 95
  SEQ External Cues - Week 6 | 70.64 (26.92)
Statistical Analysis 1: Comparison: Smiling Instead of Smoking (SiS) App Version 2; SEQ-12 - Internal; Test type: Superiority; p < .0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 13.1, 95% CI 2-sided [7.6 to 18.7]
Statistical Analysis 2: Comparison: Smiling Instead of Smoking (SiS) App Version 2; SEQ-12 - External; Test type: Superiority; p < .0001, t-test, 2 sided; Mean Difference (Final Values) = 11.1, 95% CI 2-sided [6.1 to 16.1]

8. Secondary Outcome: Within-person Changes in Theorized Mechanism of Behavior Change - Single-item Self-efficacy Measure
Description: The single-item self-efficacy measure asked: "How CONFIDENT are you that you will be able to quit smoking/stay quit?" This item was measured on a slider scale ranging from 0="not at all" to 100="extremely confident", so that higher scores indicate greater confidence in the ability to quit smoking or stay quit.
Time Frame: Baseline, 2-weeks, and 6-weeks post-quit
Population: n=1 had incomplete baseline data, n=4 were missing Week 2 data, n=5 were missing Week 6 data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
Number analyzed (Participants) | 99
units on a scale
  Baseline | 75.71 (20.05)
  2-week: number analyzed (Participants) | 96
  2-week | 76.91 (19.42)
  6-week: number analyzed (Participants) | 95
  6-week | 81.22 (22.16)
Statistical Analysis 1: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority; p = 0.0126, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 5.5, 95% CI 2-sided [1.2 to 9.8]

9. Secondary Outcome: Within-person Changes in Theorized Mechanism of Behavior Change - Single-item Motivation to Quit Measure
Description: The single-item self-efficacy measure asked: "How MOTIVATED are you to quit smoking/ stay quit?" This item was measured on a slider scale ranging from 0="not at all" to 100="extremely motivated", where higher scores indicate a greater motivation to quit smoking or stay quit.
Time Frame: Baseline, 2-weeks, and 6-weeks post-quit
Population: n=4 were missing Week 2 data, n=5 were missing Week 6 data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
Number analyzed (Participants) | 100
units on a scale
  Baseline | 88.04 (14.57)
  2-week: number analyzed (Participants) | 96
  2-week | 83.74 (18.36)
  6-week: number analyzed (Participants) | 95
  6-week | 81.73 (22.61)
Statistical Analysis 1: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority; p = 0.0053, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -6.6, 95% CI 2-sided [-11.1 to -2.0]

10. Secondary Outcome: Within-person Changes in Theorized Mechanism of Behavior Change - Attitudes Towards Smoking Scale (Etter et al., 2000)
Description: The 18-item Attitudes Towards Smoking (ATS-18) scale measures attitudes towards smoking in current and former cigarette smokers. It was rated on a 5-point Likert scale, from 1="strongly disagree" to 5="strongly agree.". The ATS-18 has 3 sub-scales: Adverse effects of smoking (items 1-10), psychoactive benefits of smoking (items 11-14), and pleasure of smoking (items 15-18). To score, all items per sub-scale were averaged to obtain a mean score within each sub-scale. For each sub-scale, higher scores indicate greater agreement with the specific attitude towards smoking.
Time Frame: Baseline, 2-weeks, and 6-weeks post-quit
Population: n=1 had incomplete baseline data, n=4 were missing Week 2 data, n=5 were missing Week 6 data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
Number analyzed (Participants) | 100
units on a scale
  ATS-18 Adverse effects of smoking - Baseline | 4.42 (0.54)
  ATS-18 Adverse effects of smoking - Week 2: number analyzed (Participants) | 96
  ATS-18 Adverse effects of smoking - Week 2 | 4.46 (0.55)
  ATS-18 Adverse effects of smoking - Week 6: number analyzed (Participants) | 95
  ATS-18 Adverse effects of smoking - Week 6 | 4.44 (0.83)
  ATS-18 Psychoactive benefits of smoking - Baseline | 3.97 (0.73)
  ATS-18 Psychoactive benefits of smoking - Week 2: number analyzed (Participants) | 96
  ATS-18 Psychoactive benefits of smoking - Week 2 | 3.59 (1.01)
  ATS-18 Psychoactive benefits of smoking - Week 6: number analyzed (Participants) | 95
  ATS-18 Psychoactive benefits of smoking - Week 6 | 3.17 (1.29)
  ATS-18 Pleasure of smoking - Baseline | 3.27 (1.00)
  ATS-18 Pleasure of smoking - Week 2: number analyzed (Participants) | 96
  ATS-18 Pleasure of smoking - Week 2 | 2.95 (1.23)
  ATS-18 Pleasure of smoking - Week 6: number analyzed (Participants) | 95
  ATS-18 Pleasure of smoking - Week 6 | 2.67 (1.29)
Statistical Analysis 1: Comparison: Smiling Instead of Smoking (SiS) App Version 2; ATS - Adverse Effects; Test type: Superiority; p = 0.76, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.1 to 0.2]
Statistical Analysis 2: Comparison: Smiling Instead of Smoking (SiS) App Version 2; ATS - Psychoactive Benefits; Test type: Superiority; p < .0001, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.0 to -0.5]
Statistical Analysis 3: Comparison: Smiling Instead of Smoking (SiS) App Version 2; ATS - Pleasure; Test type: Superiority; p < .0001, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-0.8 to -0.3]

11. Secondary Outcome: Within-person Changes in Theorized Mechanism of Behavior Change - Commitment to Quitting Scale (Kahler et al., 2007)
Description: The Commitment to Quitting Smoking Scale (CQSS) asks participants to rate their level of agreement (Likert scale, 1="strongly disagree" to 5="strongly agree") on 8-items assessing motivation to quit smoking (e.g., I'm not going to let anything get in the way of my quitting smoking).
  Scale scores are reported as the average of all items, where higher scores indicate a greater commitment to quitting smoking.
Time Frame: Baseline, 2-weeks, and 6-weeks post-quit
Population: n=1 had incomplete baseline data, n=4 were missing Week 2 data, n=5 were missing Week 6 data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
Number analyzed (Participants) | 100
units on a scale
  Baseline | 4.08 (0.67)
  Week 2: number analyzed (Participants) | 96
  Week 2 | 3.98 (0.76)
  Week 6: number analyzed (Participants) | 95
  Week 6 | 4 (0.99)
Statistical Analysis 1: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority; p = 0.25, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.1]

12. Secondary Outcome: Within-person Changes in Theorized Mechanism of Behavior Change - Decisional Balance Inventory (DBI) for Smoking Short Form (Ward et al., 2004)
Description: This 6-item form assesses the personal importance people place on positive and negative smoking expectancies. Items were rated on slider scales ranging from 0="not at all important" to 100="extremely important." Two sub-scale mean scores were calculated: positive expectancies (3 items), and negative smoking expectancies (3 items). On both scales, higher scores indicate a greater importance of the smoking expectancies (positive or negative).
Time Frame: Baseline, 2-weeks, and 6-weeks post-quit
Population: n=4 were missing Week 2 data, n=5 were missing Week 6 data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
Number analyzed (Participants) | 100
units on a scale
  DBI positive expectancies - Baseline | 56.59 (19.89)
  DBI positive expectancies - Week 2: number analyzed (Participants) | 96
  DBI positive expectancies - Week 2 | 45.01 (23.96)
  DBI positive expectancies - Week 6: number analyzed (Participants) | 95
  DBI positive expectancies - Week 6 | 35.97 (29.49)
  DBI negative expectancies - Baseline | 68.61 (26.24)
  DBI negative expectancies - Week 2: number analyzed (Participants) | 96
  DBI negative expectancies - Week 2 | 66.44 (26.25)
  DBI negative expectancies - Week 6: number analyzed (Participants) | 95
  DBI negative expectancies - Week 6 | 66.17 (28.93)
Statistical Analysis 1: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — DBI - Positive Experiences; p < .0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -20.7, 95% CI 2-sided [-27.2 to -14.3]
Statistical Analysis 2: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — DBI - Negative Experiences; p = 0.27, t-test, 2 sided — We used hierarchical linear mixed models with maximum likelihood estimation to handle missing data, then used a planned, pairwise comparison to test for within-person changes between baseline and week 6."; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-8.1 to 2.3]

13. Secondary Outcome: Within-person Changes in Theorized Mechanism of Behavior Change - Single-item Pros/Cons of Quitting Smoking Measures
Description: Two single-item measures assessed the pros and cons of being smoke-free: (1) "Think about all the things you LIKE/LOVE about quitting/being smoke-free; taken together, how important are those things to you RIGHT NOW?" and (2) "Think about all the things you DISLIKE/HATE about quitting/being smoke-free; taken together, how important are those things to you RIGHT NOW?" Both single-item measures were rated on slider scales ranging from 0="not at all" to 100="extremely important", so that higher scores indicate a greater perceived importance of the pros and cons of being smoke-free, respectively.
Time Frame: Baseline, 2-weeks, and 6-weeks post-quit
Population: n=4 and n=5 participants had missing data at weeks 2 and 6, respectively. Data was analyzed in a hierarchical mixed model with maximum likelihood estimation to handle missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
Number analyzed (Participants) | 100
units on a scale
  Pros of being smoke-free - Baseline | 84.90 (21.12)
  Pros of being smoke-free - Week 2: number analyzed (Participants) | 96
  Pros of being smoke-free - Week 2 | 80.40 (25.16)
  Pros of being smoke-free - Week 6: number analyzed (Participants) | 95
  Pros of being smoke-free - Week 6 | 75.71 (31.01)
  Cons of being smoke-free - Baseline | 63.40 (32.25)
  Cons of being smoke-free - Week 2: number analyzed (Participants) | 96
  Cons of being smoke-free - Week 2 | 64.40 (31.44)
  Cons of being smoke-free - Week 6: number analyzed (Participants) | 95
  Cons of being smoke-free - Week 6 | 58.51 (35.80)
Statistical Analysis 1: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — Pros of Being Smoke-Free; p = 0.009, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -9.1, 95% CI 2-sided [-15.9 to -2.3]
Statistical Analysis 2: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — Cons of Quitting; p = 0.25, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -5.1, 95% CI 2-sided [-13.7 to 3.6]

14. Secondary Outcome: Within-person Changes in Theorized Mechanism of Behavior Change - Perceived Stress Scale (PSS) (Cohen, 1983)
Description: This 10-item scale assesses perceived stress during the past month. Items were rated on a 5-point Likert scale ranging from 0="Never" to 4="Very Often." The overall scale score is the total of all 10 items, of which 4 are reverse-coded, so that score totals can range from 0 to 40 with higher scores indicating greater levels of perceived stress. The PSS has two sub-scales that assess perceived helplessness (6 items) and perceived self-efficacy (4 items). Sub-scale scores were calculated as mean scores of all sub-scale items (sub-scale score ranges: 0-4), so that higher scores on the sub-scales indicate higher perceived helplessness or higher perceived self-efficacy, respectively.
Time Frame: Baseline, 2-weeks, and 6-weeks post-quit
Population: n=4 were missing Week 2 data, n=5 were missing Week 6 data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
Number analyzed (Participants) | 100
score on a scale
  PSS total scores - Baseline | 19.26 (7.51)
  PSS total scores - Week 2: number analyzed (Participants) | 96
  PSS total scores - Week 2 | 17.46 (7.39)
  PSS total scores - Week 6: number analyzed (Participants) | 95
  PSS total scores - Week 6 | 16.77 (8.66)
  PSS Perceived helplessness - Baseline | 2.10 (0.93)
  PSS Perceived helplessness - Week 2: number analyzed (Participants) | 96
  PSS Perceived helplessness - Week 2 | 1.93 (0.92)
  PSS Perceived helplessness - Week 6: number analyzed (Participants) | 95
  PSS Perceived helplessness - Week 6 | 1.78 (1.03)
  PSS Perceived self-efficacy - Baseline | 2.34 (0.85)
  PSS Perceived self-efficacy - Week 2: number analyzed (Participants) | 96
  PSS Perceived self-efficacy - Week 2 | 2.53 (0.80)
  PSS Perceived self-efficacy - Week 6: number analyzed (Participants) | 95
  PSS Perceived self-efficacy - Week 6 | 2.48 (0.94)
Statistical Analysis 1: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — PSS total scores; p = 0.0069, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-4.1 to -0.7]
Statistical Analysis 2: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — PSS - Perceived Helplessness; p = 0.0043, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to -0.1]
Statistical Analysis 3: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — PSS - Perceived Self-Efficacy; p = 0.1953, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.4]

15. Secondary Outcome: Within-person Changes in Theorized Mechanism of Behavior Change - Brief Coping Orientation to Problems Experienced (Carver, 1997)
Description: This 28-item scale assesses the use of 14 coping mechanisms. Each item was rated on a 4-point Likert-scale, where 1="I haven't been doing this at all", 2="I've been doing this a little bit", 3="I've been doing this a medium amount", and 4="I've been doing this a lot." Sub-scales consist of 2 items for each of 14 coping mechanisms with no reversals of coding: (1) Self-distraction, (2) active coping, (3) denial, (4) substance use, (5) use of emotional support, (6) use of instrumental support, (7) behavioral disengagement, (8) venting, (9) positive reframing, (10) planning, (11) humor, (12) acceptance, (13) religion, (14) self-blame. Sub-scale scores range from 2 to 8 with higher scores indicating more frequent use of each specific coping mechanism, regardless of whether they are considered adaptive or maladaptive.
Time Frame: Baseline, 2-weeks, and 6-weeks post-quit
Population: n=1 had incomplete baseline data for Brief COPE - Acceptance and Brief COPE denial - Baseline, n=4 were missing Week 2 data (with n=5 incomplete for Brief COPE use of emotional support, Brief COPE use of instrumental support, Brief COPE planning, Brief COPE self-blame), n=5 has incomplete baseline date (with n=6 incomplete for Brief COPE religion, Brief COPE active coping, Brief COPE Self-distraction).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
Number analyzed (Participants) | 100
score on a scale
  Brief COPE Self-distraction - Baseline | 5.91 (1.52)
  Brief COPE Self-distraction - Week 2: number analyzed (Participants) | 96
  Brief COPE Self-distraction - Week 2 | 6.46 (1.61)
  Brief COPE Self-distraction - Week 6: number analyzed (Participants) | 94
  Brief COPE Self-distraction - Week 6 | 6.28 (1.69)
  Brief COPE active coping - Baseline | 6.57 (1.22)
  Brief COPE active coping - Week 2: number analyzed (Participants) | 96
  Brief COPE active coping - Week 2 | 6.46 (1.44)
  Brief COPE active coping - Week 6: number analyzed (Participants) | 94
  Brief COPE active coping - Week 6 | 6.36 (1.61)
  Brief COPE denial - Baseline: number analyzed (Participants) | 99
  Brief COPE denial - Baseline | 3.33 (1.77)
  Brief COPE denial - Week 2: number analyzed (Participants) | 96
  Brief COPE denial - Week 2 | 3.48 (1.82)
  Brief COPE denial - Week 6: number analyzed (Participants) | 95
  Brief COPE denial - Week 6 | 3.33 (1.81)
  Brief COPE substance use - Baseline | 3.21 (1.91)
  Brief COPE substance use - Week 2: number analyzed (Participants) | 96
  Brief COPE substance use - Week 2 | 3.16 (1.88)
  Brief COPE substance use - Week 6: number analyzed (Participants) | 95
  Brief COPE substance use - Week 6 | 3.12 (1.86)
  Brief COPE use of emotional support - Baseline | 5.12 (1.85)
  Brief COPE use of emotional support - Week 2: number analyzed (Participants) | 95
  Brief COPE use of emotional support - Week 2 | 5.68 (1.93)
  Brief COPE use of emotional support - Week 6: number analyzed (Participants) | 95
  Brief COPE use of emotional support - Week 6 | 5.40 (2.02)
  Brief COPE use of instrumental support - Baseline | 5.35 (1.98)
  Brief COPE use of instrumental support - Week 2: number analyzed (Participants) | 95
  Brief COPE use of instrumental support - Week 2 | 5.44 (1.88)
  Brief COPE use of instrumental support - Week 6: number analyzed (Participants) | 95
  Brief COPE use of instrumental support - Week 6 | 5.46 (1.93)
  Brief COPE behavioral disengagement - Baseline | 3.26 (1.42)
  Brief COPE behavioral disengagement - Week 2: number analyzed (Participants) | 96
  Brief COPE behavioral disengagement - Week 2 | 3.28 (1.71)
  Brief COPE behavioral disengagement - Week 6: number analyzed (Participants) | 95
  Brief COPE behavioral disengagement - Week 6 | 3.52 (1.79)
  Brief COPE venting - Baseline | 5.13 (1.67)
  Brief COPE venting - Week 2: number analyzed (Participants) | 96
  Brief COPE venting - Week 2 | 4.96 (1.84)
  Brief COPE venting - Week 6: number analyzed (Participants) | 95
  Brief COPE venting - Week 6 | 4.60 (1.85)
  Brief COPE positive reframing - Baseline | 6.10 (1.62)
  Brief COPE positive reframing - Week 2: number analyzed (Participants) | 96
  Brief COPE positive reframing - Week 2 | 6.22 (1.62)
  Brief COPE positive reframing - Week 6: number analyzed (Participants) | 95
  Brief COPE positive reframing - Week 6 | 5.87 (1.85)
  Brief COPE planning - Baseline | 6.55 (1.40)
  Brief COPE planning - Week 2: number analyzed (Participants) | 95
  Brief COPE planning - Week 2 | 6.12 (1.76)
  Brief COPE planning - Week 6: number analyzed (Participants) | 95
  Brief COPE planning - Week 6 | 5.95 (1.76)
  Brief COPE humor - Baseline | 4.48 (2.00)
  Brief COPE humor - Week 2: number analyzed (Participants) | 96
  Brief COPE humor - Week 2 | 4.35 (2.12)
  Brief COPE humor - Week 6: number analyzed (Participants) | 95
  Brief COPE humor - Week 6 | 4.42 (2.09)
  Brief COPE acceptance - Baseline: number analyzed (Participants) | 99
  Brief COPE acceptance - Baseline | 5.76 (1.48)
  Brief COPE acceptance - Week 2: number analyzed (Participants) | 96
  Brief COPE acceptance - Week 2 | 6.23 (1.52)
  Brief COPE acceptance - Week 6: number analyzed (Participants) | 95
  Brief COPE acceptance - Week 6 | 6.20 (1.69)
  Brief COPE religion - Baseline | 4.37 (2.14)
  Brief COPE religion - Week 2: number analyzed (Participants) | 96
  Brief COPE religion - Week 2 | 4.51 (2.29)
  Brief COPE religion - Week 6: number analyzed (Participants) | 94
  Brief COPE religion - Week 6 | 4.56 (2.31)
  Brief COPE self-blame - Baseline | 4.79 (2.07)
  Brief COPE self-blame - Week 2: number analyzed (Participants) | 95
  Brief COPE self-blame - Week 2 | 4.09 (1.86)
  Brief COPE self-blame - Week 6: number analyzed (Participants) | 95
  Brief COPE self-blame - Week 6 | 3.99 (2.13)
Statistical Analysis 1: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — Brief COPE Self-distraction; p = 0.087, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.1 to 0.8]
Statistical Analysis 2: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — Brief COPE active coping; p = 0.2866, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.209, 95% CI 2-sided [-0.6 to 0.2]
Statistical Analysis 3: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — Brief COPE denial; p = 0.9296, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.4 to 0.4]
Statistical Analysis 4: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — Brief COPE substance use; p = 0.6599, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.5 to 0.3]
Statistical Analysis 5: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — Brief COPE use of emotional support; p = 0.2315, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.2 to 0.7]
Statistical Analysis 6: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — Brief COPE use of instrumental support; p = 0.6183, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.3 to 0.6]
Statistical Analysis 7: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — Brief COPE behavioral disengagement; p = 0.2037, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.1 to 0.7]
Statistical Analysis 8: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — Brief COPE venting; p = 0.0060, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.9 to -0.2]
Statistical Analysis 9: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — Brief COPE positive reframing; p = 0.3045, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.7 to 0.2]
Statistical Analysis 10: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — Brief COPE planning; p = 0.0029, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.0 to -0.2]
Statistical Analysis 11: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — Brief COPE humor; p = 0.8274, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.5 to 0.4]
Statistical Analysis 12: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — Brief COPE acceptance; p = 0.0349, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [0.0 to 0.9]
Statistical Analysis 13: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — Brief COPE religion; p = 0.3451, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.6]
Statistical Analysis 14: Comparison: Smiling Instead of Smoking (SiS) App Version 2; Test type: Superiority — Brief COPE self-blame; p = 0.0006, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.2 to -0.3]

16. Other Pre Specified Outcome: Features of App That Need Improvement - App Usage
Description: App usage, as quantified by the number of days of used during the prescribed period of app use (i.e., 49), based on passively recorded app usage patterns.
Time Frame: 6 weeks after chosen smoking cessation date
Measure: Mean (Standard Deviation); unit: days on which app was used at least once
Arm/Group | Smiling Instead of Smoking App
Number analyzed (Participants) | 100
days on which app was used at least once | 24.7 (13.8)

17. Other Pre Specified Outcome: Self-reported Smoking Status
Description: Participants were asked "Have you been abstinent during the past 30 days?" in follow-up to providing their current smoking status as "I do not smoke at all." The outcome is presented as a % of participants who self-reported 30-day point-prevalence smoking abstinence. Participants were assumed to be smoking if they did not complete surveys.
Time Frame: Baseline, 2 weeks post-quit, 6 weeks post-quit, 3-months post-quit, 6-months post-quit
Measure: Count of Participants; unit: Participants
Arm/Group | Smiling Instead of Smoking App
Number analyzed (Participants) | 100
Participants
  Baseline | 0
  2 weeks post-quit | 1
  6 weeks post-quit | 40
  3-months post-quit | 56
  6-months post-quit | 56

ADVERSE EVENTS:
Time Frame: Baseline to 6-month post-quit follow-up
Description: No participant reported any adverse event.
Arm/Group | Smiling Instead of Smoking (SiS) App Version 2
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT03951766/Prot_SAP_ICF_000.pdf